CLINICAL TRIAL: NCT00054340
Title: Conditioning With Targeted Busulfan, Cyclophosphamide and Thymoglobulin for Allogeneic Marrow or Peripheral Blood Stem Cell (PBSC) Transplantation for Myelodysplasia and Myeloproliferative Disorders
Brief Title: Combination Chemotherapy and Antithymocyte Globulin in Reducing Graft-Versus-Host Disease in Patients Undergoing Donor Stem Cell Transplantation For Myelodysplastic Syndrome or Myeloproliferative Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Supportive Care
Other Study IDs: 1723.00; FHCRC-1723.00; CDR0000270397 (Registry Identifier: PDQ)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: graft versus host disease; polycythemia vera; chronic idiopathic myelofibrosis; essential thrombocythemia; untreated adult acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; chronic eosinophilic leukemia; chronic neutrophilic leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Myeloid, Acute; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Congenital Abnormalities | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Cyclosporine; Methotrexate; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Combining antithymocyte globulin with combination chemotherapy before donor peripheral stem cell transplantation may reduce the chance of developing graft-versus-host disease following transplantation.

PURPOSE: Phase I/II trial to study the effectiveness of combining antithymocyte globulin with busulfan and cyclophosphamide in reducing graft-versus-host disease in patients who are undergoing donor stem cell transplantation for myelodysplastic syndrome or other myeloproliferative disorder.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence of acute graft-vs-host disease (GVHD) requiring therapy in patients with myelodysplastic syndromes or myeloproliferative disorders treated with busulfan, cyclophosphamide, and anti-thymocyte globulin prior to transplantation with filgrastim (G-CSF)-mobilized peripheral blood stem cells (or bone marrow) from related or unrelated donors.
* Determine the incidence of relapse and relapse-free survival in patients treated with this regimen.
* Determine the incidence of non-relapse mortality by day 100 and 1 year posttransplantation in patients treated with this regimen.
* Determine the incidence of Epstein-Barr virus reactivation, infections, and chronic GVHD in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of anti-thymocyte globulin.

* Conditioning and graft-vs-host disease (GVHD) prophylaxis: Patients receive oral busulfan every 6 hours on days -7 to -4 (16 doses), cyclophosphamide IV on days -3 and -2, and anti-thymocyte globulin IV over 3 hours on days -3, -2, and -1.

Cohorts of 15 patients receive adjusted doses of anti-thymocyte globulin to determine the optimal dose at which Epstein-Barr virus (EBV) activation and GVHD are reduced. The optimal dose is the dose at which 2 consecutive cohorts receive the same regimen.

* Stem cell transplantation: Patients undergo peripheral blood stem cell (PBSC) or bone marrow transplantation on day 0.
* Posttransplantation GVHD prophylaxis: Patients receive cyclosporine IV continuously on days -1 to 4 and then orally twice daily until day 180. Patients also receive methotrexate on days 1, 3, 6, and 11.

Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 30-45 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Myelodysplastic syndromes (including those that have evolved to acute myeloid leukemia)
  * Myeloproliferative disorders

    * No chronic myelogenous leukemia
  * Other diseases eligible for conditioning with targeted busulfan, cyclophosphamide, and anti-thymocyte globulin that are not candidates for other studies
* Available related or unrelated donor compatible for HLA-A, -B, -C, DRB1, and DQB1

  * A single allele mismatch at HLA-A, -B, -C, or DRB1 is allowed

PATIENT CHARACTERISTICS:

Age

* 65 and under

Performance status

* Not specified

Life expectancy

* No severe limitation due to other diseases

Hematopoietic

* Not specified

Hepatic

* AST no greater than 2 times normal
* No hepatic disease

Renal

* Creatinine no greater than 2 times upper limit of normal OR
* Creatinine clearance at least 50% for age, gender, and weight

Cardiovascular

* No cardiac insufficiency requiring treatment
* No symptomatic coronary artery disease

Pulmonary

* No severe or mild hypoxemia

  * pO_2 at least 70 mm Hg and DLCO at least 70% of predicted OR
  * pO_2 at least 80 mm Hg and DLCO at least 60% of predicted

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No growth factors given posttransplantation concurrently with methotrexate immunosuppression

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-10; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Joachim Deeg, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States